CLINICAL TRIAL: NCT05989958
Title: A Multicenter, Randomized, Controlled, Open-Label Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability and Efficacy of HepaCure Plus DPMAS Versus DPMAS Alone in Chinese Subjects with Acute-On-Chronic Liver Failure
Brief Title: The Safety ,Tolerability and Efficacy Study of HepaCure in Chinese Subjects with Acute-On-Chronic Liver Failure
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hexaell Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCB-201
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Acute on Chronic Hepatic Failure; Liver Failure; Hepatitis
MeSH Terms: conditions — Liver Failure; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HepaCure (Experimental): Patients will receive Hepacure treatment ffollowing the treatment of DPMAS and LPE
  Interventions: Combination Product: HepaCure
- DPMAS and LPE (Active Comparator): Patients will receive DPMAS and LPE treatment
  Interventions: Device: DPMAS and LPE

INTERVENTIONS:
Combination Product: HepaCure — HepaCure will be administered in extracorporal dialysis following the treatment of DPMAS and LPE.
  Arms: HepaCure
Device: DPMAS and LPE — Using DPMAS and LPE for extracorporeal dialysis treatment.
  Arms: DPMAS and LPE

SUMMARY:
This is a multicenter, randomized, controlled, open-label phase 1/2 clinical study conducted in China to evaluate the efficacy, safety and tolerability of hiHep cell-based bio-artificial liver support system (HepaCure) plus DPMAS versus DPMAS alone in Chinese subjects with acute-on-chronic liver failure（ACLF）.

Phase 1 is a multicenter, open label study to evaluate the safety and tolerability of single dose and multiple doses of HepaCure with different treatment duration plus DPMAS in ACLF subjects respectively.

Phase 2 is a multicenter, randomized and controlled open label study to evaluate the efficacy, safety and tolerability of HepaCure plus DPMAS and LPE in ACLF subjects

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate effectively with investigators and sign the informed consent form (ICF) voluntarily.
2. Age: ≥ 18 years and ≤ 65 years.
3. Body weight: ≥ 40kg;
4. Met the criteria of ACLF in the early and middle stages in screening period (Guidelines for the Diagnosis and Treatment of Liverfilture (2018 Edition)): base on chronic liver disease, acute jaundice deepened and coagulation dysfunction caused by various inducements, manifested as extreme fatigue, with obvious gastrointestinal symptoms such as anorexia, vomiting, abdominal distention, etc; Progressive deepening of jaundice, serum TBil ≥ 171 μmol/L or increase ≥ 17.1 μmol/L daily or ≥10 × upper limit of normal value; with bleeding tendencies or manifestations (bleeding spots or ecchymosis), or 20%<PTA ≤ 40% (or 1.5 ≤ INR<2.6), and other reasons excluded.

Exclusion Criteria:

1. Subjects with primary or metastatic liver cancer.
2. Subjects with severe esophageal/gastric varices and high risk of bleeding, with positive red signs, or with previous active bleeding, as indicated by gastroscopy or imaging examination results.
3. Serum creatinine was greater than 132.6 μmol/L.
4. Subjects with serious uncontrolled infections, including sepsis, septic shock, severe pneumonia (refers to the diagnostic criteria of the American Society of Infectious Diseases/American Thoracic Society for adult severe pneumonia in 2007), abdominal infection (exist Peritonitis manifestations or white blood cells in ascites>0.1 × 10 9/L after reasonable antibiotic treatment), etc;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | From the initiation of treatment until 14 days after the end of study treatment.]
  Based on the recorded adverse events (AE), serious adverse events (SAE), adverse events of special interest (AESI), and device deficiencies (such as leakage caused by the inherent quality issues of the plasma bio-purification column), the safety from the start of the study treatment until 14 days after the end of the study treatment was evaluated.（Phase I）
survival rate | 12 weeks after the initial treatment]
  The survival rate without liver transplantation at 12 weeks after the first treatment.（PhaseⅡ） Absolute change from baseline in the MELD score of subjects at week 4 after the first treatment. （PhaseⅡ）

CONTACTS AND LOCATIONS:
Overall Officials: YU Chen, MD, Study Chair — Beijing YouAn Hospital
Locations (1):
- Beijing You'an Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China